CLINICAL TRIAL: NCT02033772
Title: Prospective Data Collection of Patients < 6 Months of Age Undergoing Thoracoscopic Surgery
Status: Completed | Type: Observational
Sponsor: Arlyne Thung (Other)
Responsible Party: Sponsor-Investigator, Arlyne Thung, Assistant Clinical Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB12-00503
Record Dates: First submitted 2013-11-22; First posted 2014-01-13 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Congenital Diaphragmatic Hernia; Tracheoesophageal Fistula; Esophageal Atresia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Tracheoesophageal Fistula; Esophageal Atresia | interventions — Thoracoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracoscopic surgery: Infants undergoing thoracoscopic surgery.
  Interventions: Procedure: Thoracoscopic surgery

INTERVENTIONS:
Procedure: Thoracoscopic surgery

SUMMARY:
The study is primarily a descriptive study examining the physiological, ventilatory, surgical, and recovery effects of patients ≤ 6 months of age who undergo thoracoscopic surgery and to determine the accuracy of transcutaneous CO2 (TC-CO2) and end-tidal CO2 (ET-CO2) during high frequency oscillatory ventilation (HFOV) and thoracoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for thoracoscopic surgery
* Patients aged ≤ 6 months of age

Exclusion Criteria:

* Patients presenting for any procedure other than thoracoscopic surgery
* Patients aged > 6 months of age

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants < 6 months of age undergoing thoracoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-08; Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Change in transcutaneous CO2 | Duration of surgery, average of 3 hours.

SECONDARY OUTCOMES:
Change in ET-CO2 | Duration of surgery, average of 3 hours.
  End-tidal CO2
Change in heart rate | Duration of surgery, average of 3 hours.
Change in blood pressure | Duration of surgery, average of 3 hours.
  Non-invasive and invasive.
Change in SpO2 | Duration of surgery, average of 3 hours.
  Oxygen saturation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States